CLINICAL TRIAL: NCT04813211
Title: Effectiveness and Safety of Mobile Artificial Cervical Vertebrae Replacement for Patients With Cervical Spondylosis: Study Protocol for a Prospective, Non-randomized Controlled, Clinical Trial
Brief Title: Effectiveness and Safety of Mobile Artificial Cervical Vertebrae Replacement for Patients With Cervical Spondylosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xi'an International Medical Center Hospital (Other)
Collaborators: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, Qiang Yin, Director, Xi'an International Medical Center Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XianInternationalMCH_HXJ_02
Record Dates: First submitted 2021-03-17; First posted 2021-03-24 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Cervical Spondylosis
Keywords: cervical spondylosis; cervical spine; intervertebral disc; joint replacement
MeSH Terms: conditions — Spondylosis | interventions — Gene Fusion; Control Groups

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two or more groups in parallel for the duration of the study
Masking Description: Nonrandomized Trial: participants are expressly assigned to intervention groups through a non-random method, such as physician choice
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trial group (Experimental): 20 patients with cervical spondylosis undergoing mobile artificial cervical vertebrae replacement
  Interventions: Procedure: mobile artificial cervical vertebrae replacement
- Control group (Experimental): 20 patients with cervical spondylosis undergoing anterior cervical corpectomy and fusion
  Interventions: Procedure: anterior cervical corpectomy and fusion

INTERVENTIONS:
Procedure: mobile artificial cervical vertebrae replacement — 1. Position: The patient is in a supine position with the neck hyperextended, ensuring his/her neck and shoulders in a stable and neutral position before surgery and the cervical spine in a "physiological" curvature position.
  2. Anesthesia: General anesthesia via oral tracheal intubation.
  3. Surgical approach: Anterior cervical spine approach through the space between the visceral sheath and the vascular sheath.
  4. Surgical method: Two intervertebral discs with adjacent lesions and part of the vertebral body between them will be removed. A curette is used to carefully strike off the annulus fibrosus and cartilage on the surface of the adjacent upper and lower endplates. Intraoperatively, the midlines of the segment and the vertebra to be replaced should be mapped out. When decompression, the midline for decompression should not be deviated from the planned midlines.
  Other Names: Trial group
  Arms: Trial group
Procedure: anterior cervical corpectomy and fusion — 1. Position: The patient is in a supine position with the neck hyperextended.
  2. Anesthesia: General anesthesia via oral tracheal intubation.
  3. Surgical approach: Anterior cervical spine approach through the space between the visceral sheath and the vascular sheath.
  4. Surgical method: Two intervertebral discs with adjacent lesions and part of the vertebrae between them will be removed. A curette will be used to carefully strike off the annulus fibrosus and cartilage on the surface of the adjacent upper and lower endplates. The removed vertebral bone will be trimmed into cancellous bone particles and filled in a cervical titanium cage with an appropriate size. The titanium cage will be implanted into the vertebral space, and fixed with adjacent vertebrae using anterior cervical titanium plates and screws.
  Other Names: Control group
  Arms: Control group

SUMMARY:
The research team designed an artificial cervical joint prosthesis suitable for subtotal resection of the lower cervical vertebral body. Previous studies regarding cadaver and animal experiments have found that this artificial joint not only retains the normal range of physiological motion of the joint, but also has good stability. Preliminary studies have shown that the designed joints are sufficiently safe and stable. The titanium materials for joints have been verified for their toxicology in long-term clinical trials and have been monitored under relevant national testing agencies in China.

DETAILED DESCRIPTION:
Artificial cervical disc technology has achieved certain clinical effects in the treatment of single-segment lesions of the lower cervical spine. However, simple artificial cervical disc replacement is only applicable for single-segment disc herniation, but not for two adjacent cervical segmental lesions, concurrent with vertebral hyperplasia and ossification of the posterior longitudinal ligament in the cervical spine. Traditional vertebral corpectomy and bone graft fusion can reduce the mobility of the cervical spine. Therefore, non-fusion fixation for such diseases has been a key issue to improve the efficacy of surgical treatments.

To this end, the research team designed an artificial cervical joint prosthesis suitable for subtotal resection of the lower cervical vertebral body. Previous studies regarding cadaver and animal experiments have found that this artificial joint not only retains the normal range of physiological motion of the joint, but also has good stability. Preliminary studies have shown that the designed joints are sufficiently safe and stable. The titanium materials for joints have been verified for their toxicology in long-term clinical trials and have been monitored under relevant national testing agencies in China.

To serve clinical patients faster and ensure that the trial design is safe, this study is designed to observe the effectiveness and safety of mobile artificial cervical vertebrae replacement for patients with cervical spondylosis.

ELIGIBILITY:
Inclusion Criteria:

* (1)Age: 18-70 years, irrespective of sex;
* (2)For mobile artificial cervical vertebrae replacement, patients with cervical spondylosis who are planned to undergo anterior cervical corpectomy and resection of two adjacent intervertebral discs;
* (3)For anterior cervical corpectomy and fusion, patients with cervical spondylosis who are planned to undergo anterior cervical corpectomy and resection of two adjacent intervertebral discs;

Exclusion Criteria:

* (1) Patients who have participated in other clinical studies 3 months before the inception of the study;
* (2) Abnormalities in liver and kidney functions (aspartate aminotransferase, alanine aminotransferase, blood creatinine and urea nitrogen levels are 1.5 times higher than normal);
* (3) Obvious abnormalities in the blood system;
* (4) Abuse of drugs or ethanol;
* (5) Patients who have brain disorders, abnormal judging ability, or cannot cooperate with the observer;
* (6) Coronary heart disease or severe kidney disease;
* (7) Severe metabolic diseases and endocrine diseases that are out of drug control;
* (8) Pregnant and lactating women and couples who are about to become pregnant in the near future;
* (9) Severe lung diseases such as asthma and lung dysfunction;
* (10) Immunodeficiency;
* (11) Single-segment intervertebral disc herniation or compression;
* (12) 3 or more vertebral segments herniated or spinal cord compression due to ligament ossification;
* (13) Active infection (systemic or local cervical spine) or a history of local cervical spine infection;
* (14) A history of anterior cervical surgery;
* (15) Patients with a need for posterior surgical treatments, with severe arthritis of the cervical spine joint process, and with spinal cord compression on the back;
* (16) Severe osteoporosis;
* (17) Cervical vertebra deformity;
* (18) A history of ossification of the posterior longitudinal ligament of the cervical spine, ankylosing spondylitis, and heterotopic ossification;
* (19) Severe cervical spine instability or trauma to the posterior structure of the cervical spine, and cervical spondylolisthesis;
* (20) Abnormal soft tissues anterior to the cervical spine (tracheal or esophageal malformations, and a history of radiotherapy), and obesity;
* (21) Allergy to prosthetic materials;
* (22) Patients who have tumors that cannot be completely resected and patients who are predicted to suffer prosthetic loosening during survival time;
* (23) Other contraindications for surgery.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Cervical joint range of motion at 6 months after operation | 6 months after operation
  Testing methods for cervical joint mobility include: Cervical joint range of motion in all directions will be accurately obtained through an in vitro infrared measurement after artificial joint replacement (joint range in °).

SECONDARY OUTCOMES:
Cervical fusion rate at 3 to 6 months after operation | 3 to 6 months after operation
  A successful fusion is assessed according to Brantigan and Steffee's imaging rating scale:
  Suspicious bone fusion: bone bridge formation in the entire fusion area with a density at least similar to postoperative data, and no light-transmitting band between the grafted bone and the vertebral body; Strong fusion: the fused bone in the fusion area is more mature and dense as shown on postoperative images. A sclerosis zone between the grafted bone and the vertebral body indicates the fusion, but there is no interface between the grafted bone and the vertebral body, and the mature bone trabecula forms a bone bridge. The bone spurs on the anterior side of the vertebral body will be absorbed, and the bone graft in the intervertebral space will move forward until the facet joints are fused. Fusion rate = (number of successfully fused patients/total number of patients) × 100% (Fusion rate in percentage).
Cervical joint range of motion at 7 days to 3 months after operation | 3 to 6 months after operation
  Testing methods for cervical joint mobility include
  1. X-ray: The mobility of the cervical spine during flexion and extension, lateral flexion, and rotation;
  2. Coda Motion, an internationally advanced joint mobility measuring instrument of the experimental unit, will be used to measure cervical spine mobility;
  3. Cervical joint range of motion in all directions will be accurately obtained through an in vitro infrared measurement after artificial joint replacement.
Japanese Orthopaedic Association (JOA) scores at 7 days to 6 months after operation | 7 days to 6 months after operation
  JOA scoring involves upper limb motor function (4 points), lower limb motor function (4 points), sensation (6 points) and bladder function (3 points). The higher score indicates the better motor function
Neck Disability Index (NDI) scores at 7 days to 6 months after operation | 7 days to 6 months after operation
  NDI is mainly used for assessing cervical spine function. The higher score indicates the severer cervical spine dysfunction.
Visual analogue scale (VAS) scores at 7 days to 6 months after operation | 7 days to 6 months after operation
  VAS is mainly used for pain assessment. The higher score indicate the severer pain.
CT images of the cervical spine at 7 days postoperatively | 7 days after operation
  CT images of the cervical spine are used to evaluate the implantation of the artificial cervical joint.
X-ray of the cervical spine at 7 days to 6 months after operation | 7 days to 6 months after operation
  X-ray of the cervical spine is used for evaluating the morphology of the implanted cervical joint morphology.

OTHER OUTCOMES:
The incidence of adverse events at 7 days to 6 months after operation. | 7 days to 6 months after operation
  Adverse events include implant shedding, displacement, joint loosening, fracture, prolapse, infection, and heterotopic ossification. The incidence of adverse events = (number of patients with adverse events/total number of patients)×100%.

CONTACTS AND LOCATIONS:
Overall Officials: Xijing He, MD, Principal Investigator — Xi'an International Medical Center Hospital
Locations (1):
- Xi'an International Medical Center Hospital, Xi'an, Shaanxi, China